CLINICAL TRIAL: NCT03719235
Title: Accuracy of Linear Measurements of Ultra-low Dose Cone Beam Computed Tomography and Digital Panoramic Radiography Performed on Mandibular Anaesthetic Landmarks Versus Real Mandibular Measurements
Brief Title: Accuracy of Linear Measurements of Ultra-low Dose Cone Beam Computed Tomography and Digital Panoramic Radiography
Acronym: CBCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hala Wafik Mohamed El Fayoumy, principal investigator, Cairo University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HWEF
Record Dates: First submitted 2018-10-22; First posted 2018-10-25 (Actual); Last update posted 2018-10-25 (Actual); Status verified 2018-10

CONDITIONS: Cone Beam Computed Tomography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- column (Other): ultra-low dose CBCT versus digital panoramic radsiography
  Interventions: Other: CBCT

INTERVENTIONS:
Other: CBCT — ultra-low dose CBCT

SUMMARY:
measurements performed directly on dry mandibles will be compared with measurements obtained from CBCT( ultra-low dose) scans and Digital panoramic radiography.

DETAILED DESCRIPTION:
Mandibular anaesthetic landmarks will be identified on each dry mandible and will be marked using gutta percha.

The ten human dry mandibles will be submitted for:

1. Digital Panoramic Radiography. Panoramic radiographs will be obtained using the SOREDEX CRANEX™ 3Dx unit. The exposure parameters will be 8Ma, 63kVp and 16.4 sec exposure time.
2. Cone Beam Computed Tomography (CBCT). SOREDEX CRANEX™ 3Dx unit will be used in this study. Images will be acquired at a single rotation. SOREDEX® MiniDose parameters will be used. The exposure parameters will be 3.2 Ma, 90kVp and 2.3 sec exposure time to take the advantage of 3D data in dose sensitive cases like children, or reduce the radiation dose for the patient.

The real linear measurements will be measured in millimeter on dry mandibles using digital caliper and will be compared with measurements obtained from both techniques.

Images will be evaluated by two experienced radiologists of ten years of experience. Each one will evaluate the images separately twice with a period of two weeks in-between the two reading sessions. The researcher will measure out the real linear measurements on the dry mandibles using digital caliper.

ELIGIBILITY:
Inclusion Criteria:

* age 10 to 70 years
* no gender nor race predilection
* Either dentulous or edentulous are acceptable.

Exclusion Criteria:

* fractures
* pathology

Ages: 10 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-07-10 (Estimated); Study Completion 2020-09-10 (Estimated)

PRIMARY OUTCOMES:
assessment of diagnostic accuracy of linear measurements | within 2 years
  measurements made on dry mandibles will be compared with measurements obtained from CBCT scans & digital panoramic radiography

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-10-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT03719235/Prot_SAP_000.pdf